

## **Informed Consent Form**

## Internet-based intervention versus face-to-face clinical care for tinnitus: A randomized control trial

Clinical Trials registration number: NCT02665975

Principle Investigator: Eldré Beukes (eldre.beukes@anglia.ac.uk)

Ethical approval: Cambridge South Research Ethics Committee, 16/EE/0148. HRA

approval under IRAS project identification number 195565

Sponsor: Anglia Ruskin University

Grant: British Society of Audiology Applied Research Grant Fund

Clinical Sites: Norfolk and Norwich University Hospitals NHS Foundation Trust

Hinchingbrooke Health Care HNS Trust

Milton Keynes University Hospital NHS Foundation Trust

**Date of Informed consent version**: 31 May 2016



## PARTICIPATION CONSENT FORM (online)

Title of Project: Internet-based Versus Face-to-face Clinical Care for Tinnitus

IRAS identification: 195565

Thank you for your interest in taking part in this research. Before you agree to take part, please read all the information provided about the study first from the study participation sheet. If you have any questions arising, please do not hesitate to contact the researcher at email address: tinnitusuk@anglia.ac.uk or Telephone: 01223-698847

Please read the following statement and provide consent below by ticking each box. You must agree with all the statements to be eligible to take part in the study.

| I confirm that I have read and understood the participant information sheet version 3, dated 10 May, for this study. I understand what the research involves, and all my questions have been answered to my satisfaction. |
|---|
| I understand that my participation is voluntary and that I am free to withdraw from the research at any time, for any reason and without prejudice. To do so I can send a message to <a href="mailto:tinnitusuk@anglia.ac.uk">tinnitusuk@anglia.ac.uk</a> , Telephone: 01223-698847 or a message to the therapist using the encrypted conversations facility within the treatment |
| I understand that I am free to ask any questions at any time before and during the study |
| I agree to the processing of data generated by this study to be presented and shared. I understand that no personal information will be shared as confidentiality and anonymity will be maintained and the information I provide will be safeguarded. |
| I am 18 years or older and am a resident of the UK |



| I agree to provide an email address for members of the study team to communicate with me during the study. I understand that my personal details will not be used for any other purposes |
|---|
| I understand that my GP will be informed that I am participating in this study. If the need arises to contact my GP during the study, such as to request further help for difficulties with anxiety or depression, I understand that this will be discussed with me |
| e-mail address: |
| I agree to take part in the above study |

You can print a copy of this Consent Form to keep and refer to at any time.